CLINICAL TRIAL: NCT03631966
Title: Can Botulinum Toxin Injection Relieve Pain and Improve Function in Patients With Functional Popliteal Artery Entrapment Syndrome?
Brief Title: Botulinum Toxin Injection for Functional Popliteal Artery Entrapment Syndrome
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Funding withdrawn
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Michael Fredericson, Director, Stanford PM&R Sports Medicine, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 40251
Record Dates: First submitted 2017-08-08; First posted 2018-08-15 (Actual); Last update posted 2021-03-08 (Actual); Status verified 2021-03

CONDITIONS: Functional Popliteal Artery Entrapment Syndrome; Popliteal Artery Entrapment Syndrome
MeSH Terms: conditions — Popliteal Artery Entrapment Syndrome | interventions — abobotulinumtoxinA

STUDY DESIGN:
Intervention Model Description: All patient's recruited to this study will have failed prior conservative treatment, and therefore any improvements seen in symptoms from the BTX-A injection will be considered above and beyond what was provided by conservative care. As such, each patient in this study design acts as their own case control (i.e. there is no appropriate intervention and/or placebo control group for these patients).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- BTX-A injection (Experimental)
  Interventions: Drug: Dysport

INTERVENTIONS:
Drug: Dysport — BTX-A (Dysport-Ipsen Inc.) will be injected into the proximal third of the medial and lateral gastrocnemius muscles of the symptomatic leg(s). Total dose per leg will be 400 units, 200 per injection site. Injections will be performed with the aid of real-time ultrasound (Sonosite, Bothwell, WA) guidance.

SUMMARY:
Failure to adequately diagnose and treat patients with functional popliteal artery entrapment syndrome (PAES) leads to continued pain, loss of function and poor quality of life for many patients nationwide. Currently, the primary treatment for functional PAES involves muscle resection, sometimes involving large segments of muscle, which itself can lead to functional impairment. As such, a less invasive treatment for functional PAES is desirable. The focus of this work is to determine whether Botulinum toxin type A (BTX-A) injections into the gastrocnemius muscle can lessen the mechanical forces placed on the popliteal artery by the involved muscle, thereby improving symptoms caused by impaired distal blood flow.

DETAILED DESCRIPTION:
Ten (10) patients with suspected functional popliteal artery entrapment syndrome will be recruited for this study. Dr. Michael Fredericson will recruit patients from local sports medicine clinics and sports teams. Equal men and women will be recruited, between the age of 18 and 50 years. This subcategory will reduce the potential of recruiting patients with age-related confounding causes for their symptoms.

After patients have been identified as having clinical features suggestive of PAES, confirmation of the diagnosis will involve the following in accordance with standards of care: 1) Ankle-brachial index testing with provocative maneuvers (maximal passive dorsiflexion and maximal active plantarflexion, treadmill running at a slope), 2) MRI angiography with provocative maneuvers (maximal plantar and dorsiflexion).

All patients will also complete at baseline a visual analog scale (VAS) of their pain, a lower extremity functional scale (LEFS), and lower extremity ultrasound for evaluation of gastrocnemius muscle size.

Currently, treatment of functional PAES involves surgical intervention frequently involving resection of the gastrocnemius muscle. As part of this study, BTX-A will be administered to the gastrocnemius. Patients will be informed about the indications, contraindications, and adverse events associated with BTX-A injections, and they will be informed of current standard of care options, including surgical intervention. Written consent will be obtained.

Dr. Michael Fredericson will carefully inject BTX-A (Dysport-Ipsen Inc.) into the proximal third of the medial and lateral gastrocnemius muscles of the symptomatic leg(s). Total dose per leg will be 400 units, 200 per injection site. Injections will be performed with the aid of real-time ultrasound (Sonosite, Bothwell, WA) guidance.

The premise of the intervention is that hypertrophy of the gastrocnemius muscle leads to functional entrapment of the popliteal artery at the level of the popliteal fossa with provocation maneuvers or exercise. By temporarily reducing muscle tone and promoting localized atrophy through BTX-A-induced chemodenervation, this entrapment can be relieved.

The primary outcome measures for this study will be VAS scores, LEFS scores, findings of improved blood flow on ABI with provocative maneuvers, and gastrocnemius size on ultrasound.

All patient's recruited to this study will have failed prior conservative treatment, and therefore any improvements seen in symptoms from the BTX-A injection will be considered above and beyond what was provided by conservative care. As such, each patient in this study design acts as their own case control (i.e. there is no appropriate intervention and/or placebo control group for these patients).

At 1 month, 3 months and 6 months post-injection, patients will return for clinical examination, visual analog scale (VAS) score, a lower extremity functional scale (LEFS), and lower extremity ultrasound for evaluation of gastrocnemius muscle size.

ELIGIBILITY:
Inclusion Criteria:

* To participate in the intervention portion of the study, patients must have a confirmed diagnosis of functional PAES.
* Patients must report ongoing leg pain during or after physical activity at the time of intervention.
* Patients must have failed prior conservative treatment and have been experiencing exertional leg pain for > 6 months.
* Patients must be between the age of 18 and 50.

Exclusion Criteria:

Any subject will be excluded from the study if he/she has any of the following:

* History of muscle/tendon ruptures to the lower extremities
* History of a neurological disease that would affect running or jogging
* History of adverse reactions to BTX-A
* Concomitant diagnosis of exertional compartment syndrome or other cause for leg pain.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2019-10-01 (Estimated); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
VAS scores | 12 weeks
  Visual analog scale scores
Lower extremity functional scale scores | 12 weeks
  A patient-reported measure of 20 items used to evaluate the functional status in the presence of lower extremity musculoskeletal disorders

SECONDARY OUTCOMES:
VAS scores | 4 weeks, 18 weeks, and 6 months
  Visual analog scale scores
Lower extremity functional scale scores | 4 weeks, 18 weeks, and 6 months
  A patient-reported measure of 20 items used to evaluate the functional status in the presence of lower extremity musculoskeletal disorders
blood flow on ankle-brachial indices | 4 weeks, 12 weeks, and 6 months
gastrocnemius muscle size | 4 weeks, 12 weeks, and 6 months
  as measured on lower extremity ultrasound

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University, Redwood City, California, United States

IPD SHARING:
Plan to Share IPD: No